CLINICAL TRIAL: NCT04570761
Title: Effects of Auditory Brain Stimulation by "Pink Noise" on Memory Capacities in Alzheimer's Disease: Proof of Concept Study
Acronym: PINK-AD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DR200077
Record Dates: First submitted 2020-09-08; First posted 2020-09-30 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer's Disease (AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ON-Stim (Experimental): acoustic stimulation
  Interventions: Device: Dreem headband
- OFF-Stim (Sham Comparator): no acoustic stimulation
  Interventions: Device: Dreem headband

INTERVENTIONS:
Device: Dreem headband — acoustic stimulation
  Arms: ON-Stim
Device: Dreem headband — acoustic stimulation
  Arms: OFF-Stim

SUMMARY:
Alzheimer's disease (AD) is a neurodegenerative disorder affecting almost 6% of the world's population over the age of 65. This disease, in its most typical sporadic form, is characterized by an episodic memory impairment linked to a deficit in consolidation. Many studies indicate that sleep promotes this consolidation stage during the deep slow sleep stage by facilitating the transfer of information between the hippocampus and the neocortex.

A method of acoustic brain stimulation at night by pink noises has been recently developed and has shown its effectiveness in strengthening memory consolidation in healthy volunteers. Actually, there is no study observing the effect of this new stimulation method on populations with neurodegenerative pathologies, in particular in AD for which this technique could potentially become a therapeutic option.

The hypothesis is that of a strengthening of the memory consolidation capacities in subjects with AD as has been shown in healthy subjects.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a neurodegenerative disorder affecting almost 6% of the world's population over the age of 65. This disease, in its most typical sporadic form, is characterized by an episodic memory impairment linked to a deficit in consolidation. Many studies indicate that sleep promotes this consolidation stage during the deep slow sleep stage by facilitating the transfer of information between the hippocampus and the neocortex.

A method of acoustic brain stimulation at night by pink noises has been recently developed and has shown its effectiveness in strengthening memory consolidation in healthy volunteers. Actually, there is no study observing the effect of this new stimulation method on populations with neurodegenerative pathologies, in particular in AD for which this technique could potentially become a therapeutic option.

The hypothesis is that of a strengthening of the memory consolidation capacities in subjects with AD as has been shown in healthy subjects.

ELIGIBILITY:
Inclusion Criteria common to all participants:

* Age> 50 years at the inclusion
* Patient with regular sleep patterns
* Patient having given written consent
* Patient affiliated to a social security regimen

Inclusion criteria for subjects with Alzheimer's disease:

* Patient with a beginning Alzheimer's disease defined according to the criteria of the National Institute on Aging-Alzheimer's Association or carriers of a prodromal Alzheimer's disease defined according to the criteria of the International Working Group IWG-2; the diagnosis must be supported by brain imaging and a blood test carried out in routine care
* MMSE score ≥ 24

Inclusion criteria for healthy volunteers:

* Absence of neurodegenerative pathologies
* Matched in age (+/- 5 years) and in sex with a patient

Non-inclusion criteria common to all participants:

* Psychiatric pathologies (except depression or anxiety disorders stabilized for more than 3 months)
* History of pathology which may have consequences on cognitive functioning and / or sleep: brain tumor, constituted stroke, epilepsy, head trauma (with clinical or parenchymal sequelae objectified on brain imagery), brain surgery
* Any significant comorbidity likely to constitute a confounding factor according to the clinician
* Psychotropic treatments introduced or modified <3 months before inclusion
* Hypnotic and / or sedative treatments
* Chronic consumption of alcohol or drugs
* Legal incapacity and / or other circumstance rendering the patient unable to understand the nature, objective or consequences of the study
* Major under guardianship or curatorship
* Patient not French-speaking by birth or illiterate

Exclusion Criteria common to all participants:

* Sleep disorders defined by a score> 5 on the Pittsburg sleep quality index (PSQI)
* A score> 10 on the Epworth sleepiness index

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching. | Day 7
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching.
difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching. | Day 8
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching.
difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching. | Day 14
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching.
difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching. | Day 15
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the memory task of word matching.

SECONDARY OUTCOMES:
Number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task. | Day 7
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task.
Number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task. | Day 8
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task.
Number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task. | Day 14
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task.
Number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task. | Day 15
  gross variation of the difference between morning and eve of the number of reminders found between the "ON-stimulation" condition and the "OFF-stimulation" condition, on the ecological memory task.
The memory complaint for Mc Nair's Questionnaire | Baseline
  score from 0 to 156.156 control of a bad score. The variation between J0 and J15 will be studied.
Psychoaffective aspects (Depression) for MADRS (Montgomery Asberg Depression Rating Scale) | Baseline
  score from 0 to 60.60 control of a bad score. The variation between J0 and J15 will be studied.
Psychoaffective aspects (Anxiety) for HAMA (Hamilton Anxiety) | Baseline
  score from 0 to 56.56 control of a bad score. The variation between J0 and J15 will be studied.
Quality of sleep for Pittsburgh Index (PSQI) | Baseline
  It is more an index of tolerance than efficiency. If the score is higher, the tolerance is lower.
The memory complaint for Mc Nair's Questionnaire | Day 15
  score from 0 to 156.156 control of a bad score. The variation between J0 and J15 will be studied.
Psychoaffective aspects (Depression) for MADRS (Montgomery Asberg Depression Rating Scale) | Day 15
  score from 0 to 60.60 control of a bad score. The variation between J0 and J15 will be studied.
Psychoaffective aspects (Anxiety) for HAMA (Hamilton Anxiety) | Day 15
  score from 0 to 56.56 control of a bad score. The variation between J0 and J15 will be studied.
Quality of sleep for Pittsburgh Index (PSQI) | Day 15
  It is more an index of tolerance than efficiency. If the score is higher, the tolerance is lower.
amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition | Day 7
  gross variation in the amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition, on an ambulatory EEG device
amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition | Day 8
  gross variation in the amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition, on an ambulatory EEG device
amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition | Day 14
  gross variation in the amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition, on an ambulatory EEG device
amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition | Day 15
  gross variation in the amplitude of slow waves in deep slow sleep between the "ON-stimulation" condition and the "OFF-stimulation" condition, on an ambulatory EEG device

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tours, Tours, France